CLINICAL TRIAL: NCT02182726
Title: COX-2 Postmarketing Surveillance Study With MOBEC® 15 mg Tablets
Brief Title: Postmarketing Surveillance Study With MOBEC®
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 107.245
Record Dates: First submitted 2014-07-03; First posted 2014-07-08 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Meloxicam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- MOBEC
  Interventions: Drug: MOBEC

INTERVENTIONS:
Drug: MOBEC

SUMMARY:
The aim of the study is to investigate

* the indication for MOBEC in a dose of 15 mg per day
* the treatments patients were receiving before switching to 15 mg MOBEC
* how treatment with 15 mg is assessed compared with previous treatment
* how effective and safe treatment with 15 mg MOBEC is considered

ELIGIBILITY:
Inclusion Criteria:

* An indication for a treatment with 15 mg MOBEC of at least four weeks

  * the symptomatic short-term treatment of osteoarthritis
  * the symptomatic long-term treatment of rheumatoid arthritis (chronic polyarthritis); restriction: the recommended dose for long-term treatment of elderly patients is 7.5 mg)
  * the symptomatic treatment of ankylosing spondylitis

Exclusion Criteria:

* Treatment with MOBEC prior to the start of the study
* Patients with any of the general or specific contraindications of MOBEC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primarily internal and general medical practices
Sampling Method: Non-Probability Sample
Enrollment: 4760 (Actual)
Dates: Start 2001-05; Primary Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Nature and incidence of adverse drug reactions (ADR) | up to week 8
Assessment of efficacy by physician on a 5-point scale | up to week 8
Assessment of tolerability by physician on a 5-point scale | up to week 8